CLINICAL TRIAL: NCT01532661
Title: National Registry of rFVIIa (Novoseven) in Haemorrhagic Traumatology
Acronym: NOVO7
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Novo Nordisk A/S (Industry); Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 07 20
Record Dates: First submitted 2011-12-12; First posted 2012-02-14 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Hemorrhage; Bleeding
Keywords: TRAUMA; HAEMORRHAGIC; rVIIa; Complication of Trauma hemorrhage; bleeding; rFVIIa administration for hemorrhage after trauma
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observational study: haemorrhagic trauma received rFVIIa
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — data collected by investigators

SUMMARY:
The rFVIIa (Novoseven) has been tested in traumatic hemorrhage but its efficiency has not been proven yet in this context. A national register has been set up in France identifying the patients which received rFVIIa.

Those patients had persistent and active bleeding after severe trauma despite surgery and/or interventional radiology embolization.

The aim of this present study is to report the first clinical results in those situations of patients treated with rFVIIa.

DETAILED DESCRIPTION:
It consists of a study of a prospective cohort in 36 centers, for 3 years, from April 1st 2008. The data of all patients who received rFVIIa in traumatic situation were collected. The investigators colligated clinical and biological parameters; have been analyzed treatment received during initial care, in intensive care before and after they received rFVIIa, length of stay in ICU, secondary effects, complications and patients outcome.

ISS and TRISS score were calculated to predict mortality.

ELIGIBILITY:
Inclusion Criteria:

* people affiliated to social security
* patients admitted in ISU for haemorrhagic trauma
* patients received rFVIIa after the other treatment for bleeding control

Exclusion Criteria:

* allergy or hypersensitivity to rVIIa or one of its component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in ICU after massive bleeding trauma and received rFVIIa
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
use of rFVIIa in haemorrhagic trauma compared to guidelines | twenty four hours
  Deviations with European guidelines use of rFVIIa

SECONDARY OUTCOMES:
medico economic evaluation | one year
  number of patients receiving rFVIIa by year and posology by patient
security and efficiency use of rFVVa | thirty days
  Mandatory treatments after first dose administration of rFVIIa. Patients with serious adverse events (type) and incidence

CONTACTS AND LOCATIONS:
Overall Officials: PAYEN JF, MD, Principal Investigator — University Hospital, Grenoble
Locations (39):
- France (39):
  - MEROUANI, Alençon
  - LAIGLE, Amiens
  - SANTRE, Annecy
  - MOREL, Bordeaux
  - SEDILLOT, Bourg-en-Bresse
  - BULEON, Caen
  - MIQUET, Chambéry
  - DEBIEN, Clamart
  - GUELON, Clermont-Ferrand
  - PEASE, Clichy
  - COOK, Créteil
  - NADJI, Dijon
  - Vinsiniti, Gap
  - DECLETY, Grenoble
  - Duranteau, Le Kremlin-Bicêtre
  - GARRIGUE, Lille
  - FLOCARD, Lyon
  - GARCIN, Marseille
  - FAVIER, Metz
  - CHARBIT, Montpellier
  - YUNG, Montpellier
  - AUDIBERT, Nancy
  - CHUPIN, Nantes
  - ICHAI, Nice
  - LEFRANT, Nîmes
  - JOURNOIS, Paris
  - LANGERON, Paris
  - Mateo A Loris, Paris
  - DAVID, Pierre-Bénite
  - Nanadoumgar, Poitiers
  - LEPOUSE, Reims
  - Bleichner, Rennes
  - GUITARD, Rouen
  - MARTIN, Saint-Etienne
  - FREYS, Strasbourg
  - MEAUDRE, Toulon
  - OLIVIER, Toulouse
  - LEBAS, Vannes
  - JAULT, Villefranche-sur-Saône

REFERENCES:
- [Background] Boffard KD, Riou B, Warren B, Choong PI, Rizoli S, Rossaint R, Axelsen M, Kluger Y; NovoSeven Trauma Study Group. Recombinant factor VIIa as adjunctive therapy for bleeding control in severely injured trauma patients: two parallel randomized, placebo-controlled, double-blind clinical trials. J Trauma. 2005 Jul;59(1):8-15; discussion 15-8. doi: 10.1097/01.ta.0000171453.37949.b7. PMID 16096533
- [Result] Martinowitz U, Kenet G, Segal E, Luboshitz J, Lubetsky A, Ingerslev J, Lynn M. Recombinant activated factor VII for adjunctive hemorrhage control in trauma. J Trauma. 2001 Sep;51(3):431-8; discussion 438-9. doi: 10.1097/00005373-200109000-00002. PMID 11535886
- [Result] Rizoli SB, Boffard KD, Riou B, Warren B, Iau P, Kluger Y, Rossaint R, Tillinger M; NovoSeven Trauma Study Group. Recombinant activated factor VII as an adjunctive therapy for bleeding control in severe trauma patients with coagulopathy: subgroup analysis from two randomized trials. Crit Care. 2006;10(6):R178. doi: 10.1186/cc5133. PMID 17184516
- [Result] Harrison TD, Laskosky J, Jazaeri O, Pasquale MD, Cipolle M. "Low-dose" recombinant activated factor VII results in less blood and blood product use in traumatic hemorrhage. J Trauma. 2005 Jul;59(1):150-4. doi: 10.1097/01.ta.0000171470.39742.8e. PMID 16096555
- [Result] Delannoy B, Levrat A, Chamouard V, Aulagner G, Perdrix JP, Negrier C, Allaouchiche B. [Off label use of recombinant activated factor VII: a practice survey]. Ann Fr Anesth Reanim. 2007 Sep;26(9):774-9. doi: 10.1016/j.annfar.2007.06.001. Epub 2007 Jul 16. French. PMID 17629661